CLINICAL TRIAL: NCT04537065
Title: Refractive and Biometric Outcome Following Intravitreal Injection of Ranibizumab in Retinopathy of Prematurity: Long -Term Study
Brief Title: Long Term Outcome of Intravitreal Ranibizumab for ROP
Status: Completed | Type: Observational
Sponsor: Ameera Gamal Abdelhameed (Other)
Responsible Party: Sponsor-Investigator, Ameera Gamal Abdelhameed, Lecturer of Ophthalmology, Mansoura University
Organization: Mansoura University (Other)
Other Study IDs: Intravitreal Ranibizumab
Record Dates: First submitted 2020-08-26; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Mydriatics; Biometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- preterm infants without ROP
  Interventions: Other: cycloplegic refraction
- preterm infants with regressed ROP
  Interventions: Other: cycloplegic refraction
- preterm infants with threshold ROP
  Interventions: Other: cycloplegic refraction
- full-term infants
  Interventions: Other: cycloplegic refraction

INTERVENTIONS:
Other: cycloplegic refraction — Cycloplegic refraction and the average corneal radius of curvature were performed using a handheld auto kerato-refractometer (Righton Retinomax K-plus2). Refraction was confirmed by retinoscopy and refractive errors were calculated as spherical equivalent and astigmatism in cylinder.
  The biometric optic components, including anterior chamber depth, lens thickness, and axial length, were measured using A-scan ultrasound (model Echoscan US-4000 / 500; Nidek).
  Other Names: Biometry

SUMMARY:
premature infants who had a history of intravitreal injection of (Ranibizumab) not less than one year were examined for refractive state and biometry

DETAILED DESCRIPTION:
Medical records were collected in each group for birth history data, including gestational age (GA), birth weight (BW), and postmenstrual age (PMA) at time of intravitreal injection. The zone and stage of ROP were also recorded. All patients were evaluated for refractive errors and cycloplegic refraction was performed using a handheld auto keratorefractometer (Righton Retinomax K-plus2), and confirmed by retinoscopy examination. Refractive errors were calculated as spherical equivalent and astigmatism in cylinder. The average corneal radius of curvature was measured by handheld auto kerato-refractometer (Righton Retinomax K-plus2). The biometric optic components, including anterior chamber depth, lens thickness, and axial length, were measured using A-scan ultrasound (model Echoscan US-4000 / 500; Nidek)

ELIGIBILITY:
Inclusion Criteria:

* premature infants who had a history of intravitreal injection of (Ranibizumab) not less than one year
* Three control groups with age and sex matched were included for comparison. First group included premature infants who had ROP that regressed spontaneously without intervention. Second group was corresponded to premature infants who were diagnosed to have normal retinal vasculature from the first examination after birth. The third group belonged to full term babies

Exclusion Criteria:

* Premature infants who received intravitreal injection of (Ranibizumab) less than one year or had any ocular pathology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical records of premature infants were collected from Egyptian Neonatal Network (EGNN) data base
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
cycloplegic refraction | 1 year after injection
  Cycloplegic refraction and the average corneal radius of curvature were performed using a handheld auto kerato-refractometer (Righton Retinomax K-plus2). Refraction was confirmed by retinoscopy and refractive errors were calculated as spherical equivalent and astigmatism in cylinder
biometry | 1 year after injection
  The biometric optic components, including anterior chamber depth, lens thickness, and axial length, were measured using A-scan ultrasound (model Echoscan US-4000 / 500; Nidek). Examination under sedation was performed for uncooperative children.

CONTACTS AND LOCATIONS:
Overall Officials: Rania MR Bassiouny, MD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zin A, Gole GA. Retinopathy of prematurity-incidence today. Clin Perinatol. 2013 Jun;40(2):185-200. doi: 10.1016/j.clp.2013.02.001. PMID 23719304
- [Background] Isaza G, Arora S, Bal M, Chaudhary V. Incidence of retinopathy of prematurity and risk factors among premature infants at a neonatal intensive care unit in Canada. J Pediatr Ophthalmol Strabismus. 2013 Jan-Feb;50(1):27-32. doi: 10.3928/01913913-20121127-02. Epub 2012 Dec 4. PMID 23205771
- [Background] Lin CJ, Chen SN, Tseng CC, Chang YC, Hwang JF. Effects of ranibizumab on very low birth weight infants with stage 3 retinopathy of prematurity: A preliminary report. Taiwan Journal of Ophthalmology 2012; 2: 136-139
- [Background] Menke MN, Framme C, Nelle M, Berger MR, Sturm V, Wolf S. Intravitreal ranibizumab monotherapy to treat retinopathy of prematurity zone II, stage 3 with plus disease. BMC Ophthalmol. 2015 Mar 8;15:20. doi: 10.1186/s12886-015-0001-7. PMID 25886603
- [Background] Bassiouny, RaniaM.R. & Ellakkany, RasheedS & Aboelkhair, SamyA & Mohsen, TarekA & Othman, IhabS. (2017). Incidence and risk factors of retinopathy of prematurity in neonatal intensive care units: Mansoura, Egypt. Journal of the Egyptian Ophthalmological Society. 110. 71. 10.4103/ejos.ejos_25_17.
- [Background] Castellanos MA, Schwartz S, Garcia-Aguirre G, Quiroz-Mercado H. Short-term outcome after intravitreal ranibizumab injections for the treatment of retinopathy of prematurity. Br J Ophthalmol. 2013 Jul;97(7):816-9. doi: 10.1136/bjophthalmol-2012-302276. Epub 2012 Dec 8. PMID 23221964
- [Background] Chen YC, Chen SN, Yang BC, Lee KH, Chuang CC, Cheng CY. Refractive and Biometric Outcomes in Patients with Retinopathy of Prematurity Treated with Intravitreal Injection of Ranibizumab as Compared with Bevacizumab: A Clinical Study of Correction at Three Years of Age. J Ophthalmol. 2018 Mar 11;2018:4565216. doi: 10.1155/2018/4565216. eCollection 2018. PMID 29713524
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Cook A, White S, Batterbury M, Clark D. Ocular growth and refractive error development in premature infants with or without retinopathy of prematurity. Invest Ophthalmol Vis Sci. 2008 Dec;49(12):5199-207. doi: 10.1167/iovs.06-0114. PMID 19036998
- [Background] Dawson DG, Watsky MA, Geroski DH, Edelhauser HF. Cornea and sclera. In: Tasman W, Jaeger EA, editors. Duane's ophthalmology [CD-ROM]. Philadelphia: Lippincott Williams & Wilkins; 2007. Chapter 4